CLINICAL TRIAL: NCT06560632
Title: Phase 1 Trial of the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Clinical Activity of RP-3467 Alone and in Combination With Olaparib in Participants With Advanced Solid Tumors (POLAR Trial)
Brief Title: Phase 1 Trial of RP-3467 Alone and in Combination With Olaparib in Participants With Advanced Solid Tumors
Acronym: POLAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to terminate study early
Sponsor: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-3467-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-19 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Appointments and Schedules; olaparib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: RP-3467 monotherapy (Experimental): Eligible participants will be treated with escalating doses of RP-3467 monotherapy
  Interventions: Drug: RP-3467 at assigned dose and schedule
- Arm2: RP-3467 + Olaparib combination (Experimental): Eligible participants will be treated with escalating doses of RP-3467 in combination with Olaparib
  Interventions: Drug: RP-3467 at assigned dose and schedule; Drug: Olaparib 200-300 mg BID, daily

INTERVENTIONS:
Drug: RP-3467 at assigned dose and schedule — Eligible participants will be treated with escalating doses of RP-3467 monotherapy
Drug: Olaparib 200-300 mg BID, daily — Eligible participants will be treated with escalating doses of RP-3467 in combination with Olaparib
  Other Names: RP-3467 at assigned dose and schedule; Lynparza
  Arms: Arm2: RP-3467 + Olaparib combination

SUMMARY:
This is a multicenter, open-label Phase 1 trial to investigate the safety, PK, and pharmacodynamics of the Polθ inhibitor RP-3467 alone or in combination with the poly-ADP ribose polymerase inhibitor (PARPi) olaparib in adults with molecularly selected advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1, multi-center, open-label, dose-escalation study to:

* Evaluate the safety profile of RP-3467 when administered orally alone and in combination with olaparib and to define the MTD or MAD for RP-3467 monotherapy and the RP2D for the combination
* Characterize the PK profile of RP-3467 alone and in combination with olaparib

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years of age at the time of signing the informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant must have one of the following that has progressed or was non-responsive to prior systemic therapy and for which no standard or available known therapeutic option exists:

  1. locally advanced or metastatic epithelial ovarian cancer (including fallopian tube or primary peritoneal), or
  2. metastatic breast cancer, or
  3. metastatic castration-resistant prostate cancer (mCRPC), or
  4. pancreatic adenocarcinoma
* Measurable disease per RECIST v1.1 (exceptions for participants with non-measurable but evaluable disease [per RECIST and or PSA/CA-125])
* Next generation sequencing (NGS) report demonstrating eligible tumor biomarker
* Provision of archival tumor tissue, or if adequate archival tumor tissue is not available, provision of a fresh biopsy if there is a lesion that can be safely biopsied
* Acceptable organ function at Screening
* Acceptable hematologic function at Screening
* Life expectancy ≥12 weeks after the start of the treatment according to the Investigator's judgment

Exclusion Criteria:

* History or current condition, therapy, or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* Uncontrolled, symptomatic brain metastases.
* Presence of other known active invasive cancers
* History of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) diagnosis
* Prior therapy with a Polθ inhibitor other than RP-3467

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - # 1025, The University of California, San Francisco, California
  - # 1011, The Washington University, St Louis, Missouri
  - # 1008, Columbia University, New York, New York
  - # 1004, Memorial Sloan-Kettering Cancer Center, New York, New York
  - # 1001, The University of Texas M.D. Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 160 mg QD RP-3467: 160 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 1: 320 mg QD RP-3467: 320 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 1: 640 mg QD RP-3467: 640 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 2: 80 mg QD RP-3467 + 200 mg BID Olaparib: 80 mg RP-3467 taken QD orally in combination with 200 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
- Arm 2: 80 mg QD RP-3467 + 300 mg BID Olaparib: 80 mg RP-3467 taken QD orally in combination with 300 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
- Arm 2: 40 mg QD RP-3467 + 300 mg BID Olaparib: 40 mg RP-3467 taken QD orally in combination with 300 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
Period: Overall Study
Arm/Group | Arm 1: 160 mg QD RP-3467 | Arm 1: 320 mg QD RP-3467 | Arm 1: 640 mg QD RP-3467 | Arm 2: 80 mg QD RP-3467 + 200 mg BID Olaparib | Arm 2: 80 mg QD RP-3467 + 300 mg BID Olaparib | Arm 2: 40 mg QD RP-3467 + 300 mg BID Olaparib
Started | 1 | 3 | 4 | 3 | 2 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 4 | 3 | 2 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 160 mg QD RP-3467 | Arm 1: 320 mg QD RP-3467 | Arm 1: 640 mg QD RP-3467 | Arm 2: 80 mg QD RP-3467 + 200 mg BID Olaparib | Arm 2: 80 mg QD RP-3467 + 300 mg BID Olaparib | Arm 2: 40 mg QD RP-3467 + 300 mg BID Olaparib | Total
Number analyzed (Participants) | 1 | 3 | 4 | 3 | 2 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (0) | 55.7 (5.51) | 54.0 (13.74) | 75.0 (6.24) | 52.5 (2.12) | 55.5 (12.78) | 57.7 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 4 | 1 | 2 | 12 | 22
  Male | 1 | 0 | 0 | 2 | 0 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 1 | 3 | 3 | 2 | 2 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Any Prior PARP inhibitor therapy [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 4 | 2 | 2 | 12 | 24
  No | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experienced Dose-limiting Toxicities (DLT) During the Study Treatment
Description: The assessment of DLTs was conducted to evaluate the safety and tolerability of RP-3467 administered as monotherapy and in combination with olaparib in participants with advanced solid tumors.
Time Frame: Start of treatment to 30 days post last dose, up to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 160 mg QD RP-3467 | Arm 1: 320 mg QD RP-3467 | Arm 1: 640 mg QD RP-3467 | Arm 2: 80 mg QD RP-3467 + 200 mg BID Olaparib | Arm 2: 80 mg QD RP-3467 + 300 mg BID Olaparib | Arm 2: 40 mg QD RP-3467 + 300 mg BID Olaparib
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 1 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days post last dose, up to 13 months
Groups:
- Arm 1: 160 mg RP-3467 QD: Arm 1: 160 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 1: 320 mg RP-3467 QD: Arm 1: 320 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 1: 640 mg RP-3467 QD: Arm 1: 640 mg RP-3467 taken QD (once a day) orally in 3 weeks (21 day cycle)
- Arm 2: 80 mg RP-3467 QD+200 mg BID Ola: Arm 2: 80 mg RP-3467 taken QD orally in combination with 200 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
- Arm 2: 80 mg RP-3467 QD+300 mg BID Ola: Arm 2: 80 mg RP-3467 taken QD orally in combination with 300 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
- Arm 2: 40 mg RP-3467 QD+300 mg BID Ola: Arm 2: 40 mg RP-3467 taken QD orally in combination with 300 mg BID (twice daily) olaparib taken orally for 3 weeks (21 day cycle)
Arm/Group | Arm 1: 160 mg RP-3467 QD | Arm 1: 320 mg RP-3467 QD | Arm 1: 640 mg RP-3467 QD | Arm 2: 80 mg RP-3467 QD+200 mg BID Ola | Arm 2: 80 mg RP-3467 QD+300 mg BID Ola | Arm 2: 40 mg RP-3467 QD+300 mg BID Ola
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/4 | 0/3 | 1/2 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 1/4 | 1/3 | 1/2 | 1/13
Other Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 4/4 | 3/3 | 1/2 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 160 mg RP-3467 QD (N=1) | Arm 1: 320 mg RP-3467 QD (N=3) | Arm 1: 640 mg RP-3467 QD (N=4) | Arm 2: 80 mg RP-3467 QD+200 mg BID Ola (N=3) | Arm 2: 80 mg RP-3467 QD+300 mg BID Ola (N=2) | Arm 2: 40 mg RP-3467 QD+300 mg BID Ola (N=13)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 160 mg RP-3467 QD (N=1) | Arm 1: 320 mg RP-3467 QD (N=3) | Arm 1: 640 mg RP-3467 QD (N=4) | Arm 2: 80 mg RP-3467 QD+200 mg BID Ola (N=3) | Arm 2: 80 mg RP-3467 QD+300 mg BID Ola (N=2) | Arm 2: 40 mg RP-3467 QD+300 mg BID Ola (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders and administration site conditions) | 0 | 1 | 0 | 1 | 1 | 3
Oedema peripheral (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The Study was terminated early by the Sponsor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In this multi center study, authors are required to abide by the restriction that the first publication is to include data from all investigational sites.

DOCUMENTS (2):
  • Study Protocol (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT06560632/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT06560632/SAP_001.pdf